CLINICAL TRIAL: NCT02824770
Title: Effects of Sleep Quality on Melatonin Levels and Inflammatory Response After Major Abdominal Surgery in an Intensive Care Unit
Brief Title: Effects of Sleep Quality on Melatonin Levels and Inflammatory Response After Major Abdominal Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Eskisehir Osmangazi University (Other)
Responsible Party: Principal Investigator, Necdet Fatih Yasar, Assistant Professor, Eskisehir Osmangazi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2016-1309
Record Dates: First submitted 2016-06-28; First posted 2016-07-07 (Estimated); Last update posted 2017-06-07 (Actual); Status verified 2017-06

CONDITIONS: Sleep Deprivation
MeSH Terms: conditions — Sleep Deprivation | interventions — Bupivacaine; Tramadol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (Active Comparator): After a major abdominal surgery, the control group will receive the usual postoperative care including continous infusion of Bupivacaine (Bustesin®) via Pain Buster ® system into the wound at a rate of 5cc/hour and infusion of Tramadol HCl (Tramosel®) via PCA (Gemstar®) in the surgical intensive care unit.
  Interventions: Drug: Bupivacaine (Bustesin®) via Pain Buster ® system; Drug: Tramadol HCl (Tramosel®) via PCA system (Gemstar®); Procedure: Major abdominal surgery
- Dimming of lights and decreasing noise (Experimental): After a major abdominal surgery, the patients in the experimental group will be screened in the side-rooms where normally the patients who either have infections or are at risk of infection, are nursed and will receive continous infusion of Bupivacaine (Bustesin®) via Pain Buster ® system into the wound at a rate of 5cc/hour and infusion of Tramadol HCl (Tramosel®) via PCA (Gemstar®) as in the control group. The study intervention will include dimming of lights and decreasing noise. The lights will be dimmed to 40 lux. The doors of the side-rooms will be closed decrease the noise level below 40 dB between 11:00 p.m.-5:00 a.m.
  Interventions: Behavioral: Dimming of lights and decreasing noise level; Drug: Bupivacaine (Bustesin®) via Pain Buster ® system; Drug: Tramadol HCl (Tramosel®) via PCA system (Gemstar®); Procedure: Major abdominal surgery

INTERVENTIONS:
Behavioral: Dimming of lights and decreasing noise level — The study intervention will include dimming of lights and decreasing noise level. The lights will be dimmed to 40 lux and the doors of the side-room will be closed to decrease the noise level below 40 dB between 11:00 p.m.-5:00 a.m
  Arms: Dimming of lights and decreasing noise
Drug: Bupivacaine (Bustesin®) via Pain Buster ® system — Patients will receive continous infusion of Bupivacaine (Bustesin®) via Pain Buster ® system into the wound at a rate of 5cc/hour
Drug: Tramadol HCl (Tramosel®) via PCA system (Gemstar®) — Patients will receive infusion of Tramadol HCl (Tramosel®) via patient-controlled analgesia system (Gemstar®)
Procedure: Major abdominal surgery — Any major abdominal surgery (e.g. colectomy, gastrectomy)

SUMMARY:
Endogenous melatonin is produced by the pineal gland at night under normal conditions and regulates the sleep-wake cycle. Artificial light administered at night suppresses melatonin production and sleep disturbances are accompanied by abnormal melatonin secretion such as phase delay. Therefore, dramatic disturbances of endogenous rhythms in intensive care unit patients have remarkable effects on melatonin production. In addition to its physiological roles in regulating sleep patterns, melatonin has been demonstrated to provide antiinflammatory effects in experimental models. Although some previous studies have investigated the circadian pattern of melatonin in intensive care unit patients, the investigators think that the present study is the first one that will assess the effects of controlling noise and light on melatonin and inflammatory response after major abdominal surgery.

DETAILED DESCRIPTION:
This study is going to be conducted in accordance with the Helsinki Declaration and has been approved by Eskisehir Osmangazi University Ethics Committee. Forty consecutive patients, aged 18-65, who will undergo elective major abdominal operations will be enrolled in the study after obtaining informed consent. All patients will receive adequate postoperative pain management with the Pain Buster ® system and patient-controlled intravenous analgesia (PCA). The patients will be randomly assigned to either the experimental group or the control group. The control group will receive the usual care. The patients in the experimental group will be screened in the side-rooms where normally the patients who either have infections or are at risk of infection, are nursed. The study intervention will include dimming the lights to 40 lux and closing the doors of the side-room to decrease the noise level below 40 decibels (dB) between 11:00 p.m.-5:00 a.m.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective major abdominal surgery

Exclusion Criteria:

* Any evidence of inflammatory diseases during the postoperative care (e.g. anastomotic leakage)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-06-30 (Estimated); Study Completion 2017-07-01 (Estimated)

PRIMARY OUTCOMES:
the effect of sleep quality on the postoperative urine 6-sulphatoxymelatonin (µg - micrograms) levels | within 3 days after surgery
the effect of sleep quality on the postoperative serum c-reactive protein (mg/l - milligram/liter) levels | within 3 days after surgery
the effect of sleep quality on the postoperative serum interleukin-1 and interleukin-6 (pg/ml - picograms/milliliter) levels | within 3 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Necdet F Yasar, MD, Principal Investigator — Eskisehir Osmangazi University
Locations (1):
- Eskisehir Osmangazi University, Eskişehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Riutta A, Ylitalo P, Kaukinen S. Diurnal variation of melatonin and cortisol is maintained in non-septic intensive care patients. Intensive Care Med. 2009 Oct;35(10):1720-7. doi: 10.1007/s00134-009-1565-6. Epub 2009 Jul 4. PMID 19578832
- [Background] Hu RF, Jiang XY, Zeng YM, Chen XY, Zhang YH. Effects of earplugs and eye masks on nocturnal sleep, melatonin and cortisol in a simulated intensive care unit environment. Crit Care. 2010;14(2):R66. doi: 10.1186/cc8965. Epub 2010 Apr 18. PMID 20398302
- [Background] Seifman MA, Gomes K, Nguyen PN, Bailey M, Rosenfeld JV, Cooper DJ, Morganti-Kossmann MC. Measurement of serum melatonin in intensive care unit patients: changes in traumatic brain injury, trauma, and medical conditions. Front Neurol. 2014 Nov 17;5:237. doi: 10.3389/fneur.2014.00237. eCollection 2014. PMID 25477861